CLINICAL TRIAL: NCT05349552
Title: Safety and Efficacy of SBRT in the Treatment of Thoracic Malignant Tumors at Different Sites
Status: Recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BYSY-2022-SBRT-LC
Record Dates: First submitted 2022-04-21; First posted 2022-04-27 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Radiotherapy; Thoracic Cancer; Safety and Efficacy
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Chest Wall Type: The lesion is directly adjacent (less than 1cm) or overlapped with the chest wall.
  Interventions: Radiation: stereotactic body radiation therapy
- Peripheral Type: The lesion is more than 1cm away from the chest wall and more than 2cm away from the bronchial tree.
  Interventions: Radiation: stereotactic body radiation therapy
- Central Type: The lesion is less than 2cm away from the bronchial tree.
  Interventions: Radiation: stereotactic body radiation therapy
- Ultral-central Type: The lesion is directly adjacent or overlapped with the mediastinal structure.
  Interventions: Radiation: stereotactic body radiation therapy

INTERVENTIONS:
Radiation: stereotactic body radiation therapy — The patients were treated with high-dose and low fractionated radiotherapy, using modern precision radiotherapy technology.

SUMMARY:
SBRT (stereotactic radiotherapy) can provide a higher dose to the target area without increasing the risk of surrounding normal tissue / organ injury in selective cases. At present, SBRT has been widely used in radiotherapy of lung cancer and it can also play a better local control for lung metastasis.

However, there are parallel organs and series organs in the chest, and different organs have different tolerance to radiotherapy, so the toxicities of SBRT in different sites are different, and the prescription dose is also different.

This study intends to make a detailed division of the chest region and explore the safety and efficacy of SBRT in different areas. It is divided into four types: chest wall type: the lesion is directly adjacent or overlapped with the chest wall; peripheral type: the lesion is more than 1cm away from the chest wall and more than 2cm away from the bronchial tree; central type: the lesion is less than 2cm away from the bronchial tree; ultral-central type: the lesion is directly adjacent or overlapped with the mediastinal structure.

48-60Gy / 4-10f (EQD2 = 62.5Gy ~ 99.7Gy) was given according to the location of the tumor. Main outcome measures are local progression free survival and radiation toxicities; secondary outcome measure is overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis was malignant tumor.
* The location of the target lesion belongs to one of five types and the lesion diameter is ≤ 5cm.
* There is no extensive systemic metastasis or although there is metastasis, the metastasis have been controlled by previous treatment.
* KPS>70, no serious or uncontrolled underlying diseases, such as severe or uncontrolled hypertension, diabetes, cardiovascular and cerebrovascular diseases and organ dysfunction, and patients are expected to be tolerated by radiotherapy.

Exclusion Criteria:

* Poor basic pulmonary function or symptom correlation caused by various reasons, unable to lie flat or cooperate with treatment.
* The general condition is poor, and the expected survival time is less than 3 months.
* Psychiatric patients or poor compliance, unable to cooperate to complete treatment.
* For other reasons, the researcher believes that it is not suitable to participate in this trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chest malignant tumors who received SBRT treatment in our department from 2022 to 2025 are expected to be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Local progression free survival | From the beginning of the treatment to 2 years after the treatment.
  The time from the date of SBRT to the date of local recurrence or death or the date of last observation.
Toxicities | From the beginning of the treatment to 2 years after the treatment.
  Adverse events of radiation of normal tissues (Including lung, trachea, bronchus, esophagus, blood vessels, ribs, spinal cord, brachial plexus).

SECONDARY OUTCOMES:
Overall survival | From the beginning of the treatment to 2 years after the treatment.
  The time from the date of SBRT to the date of death from any cause or the date of last observation.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: CSR
Time Frame: Data will be available within 6 months of the study completion.
Access Criteria: Data access requests will be reviewed by an external Independent Review Panel. Requestors will be required to sign a Data Access Agreement.